CLINICAL TRIAL: NCT01748435
Title: The Role of Pre-emptive Analgesia With Qutenza (Topical Capsaicin 8%) in Preventing Neuropathic Pain Following Lower Limb Amputation: a Pilot Randomised Controlled Study
Brief Title: Pre-emptive Analgesia With Qutenza in Lower Limb Amputation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Emma Aitken, Clinical Resrach Fellow, NHS Greater Glasgow and Clyde
Other Study IDs: GU11SU387; 2012-001587-30 (EudraCT Number)
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Neuropathic Pain; Lower Limb Amputation
Keywords: Neuropathic pain; Lower limb amputation; Pre-emptive analgesia
MeSH Terms: conditions — Neuralgia | interventions — Capsaicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Qutenza: Single treatment with QUTENZA (topical capsaicin 8%) transdermal patch
  Interventions: Drug: Qutenza

INTERVENTIONS:
Drug: Qutenza — Single treatment with Qutenza
  Other Names: Qutenza (topical capsaicin 8%)

SUMMARY:
Neuropathic (nerve pain) following amputation of a limb is very common, affecting 60-80% of patients (Sherman et al, 1984). It can prolong their recovery making it difficult to fit protheses and mobilise. Current treatment options are limited and existing painkillers have significant side effects. Nevertheless there is some evidence that pre-emptive analgesia (pain relief provided prior to the surgery) has additional benefits after the surgery (Ypsilantis & Tang, 2010) Qutenza (topical capsaicin 8%)is a novel analgesic agent which is applied directly onto the skin. It works by desensitising to pain receptors in the skin (Nolano et al., 1999) and has been shown to be effective in reducing neuropathic pain in other conditions (Backonja et al., 2008) We propose to evaluate the use of Qutenza for pre-emptive analgesia in patients undergoing amputation of a limb. This is a small, pilot, randomised controlled study of 30 patients undergoing lower limb amputation who will have Qutenza or active control applied prior to surgery. They will be followed up for 12 weeks post-operatively with regular assessment of pain scores, quality of life and wound healing.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients >18 years old undergoing lower limb amputation

Exclusion Criteria:

Traumatic amputation Severe active sepsis in non-viable limb Illness necessitating urgent surgery <24 hours after admission to hospital Hypersensitivity to Qutenza, Emla or any of the excipients Broken skin or active ulceration at the site of application Severe uncontrolled hypertension (systolic BP >200) Proven cardiac event during the preceding 3 months Women who are pregnant or breast feeding Lack of capacity or inability to provide informed consent Declines participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing lower limb amputation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Chronic neuropathic pain | 12 weeks
  Chronic neuropathic pain as assessed by Visual Analogue Pain Score

SECONDARY OUTCOMES:
Neuropathic pain | 1 weeks, 6 weeks, 12 weeks
  Assessed using VAS and Brief Pain Inventory
Acute post-operative pain | Day 1, 3, 7
  Assessed by Visual Analogue Pain Score
Wound healing | 1 week
  Assessed using standardised, validated wound healing tools
Quality of life | 12 weeks
  Assessed by EQ-5D
Safety and tolerability | 1 day, 12 weeks
  Skin will be assessed for breaks/ blisters and tolerability including the need for rescue analgesia will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Emma L Aitken, MBChB, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Western Infirmary, Glasgow, Lanarkshire, United Kingdom